CLINICAL TRIAL: NCT01004328
Title: Using HIT to Improve Transitions of Complex Elderly Patients From SNF to Home
Brief Title: Using Health Information Technology (HIT) to Improve Transitions of Complex Elderly Patients From Skilled Nursing Facility (SNF) to Home
Acronym: RAMPAGEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Terry Field, Associate Professor, Meyers Primary Care Institute/University of Massachusetts Medical School., University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS017817 (AHRQ); 13001
Record Dates: First submitted 2009-07-22; First posted 2009-10-29 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Adverse Outcomes
Keywords: patient safety; care transitions; therapeutic monitoring; skilled nursing facilities; Adverse outcomes after discharge from a SNF to home

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Group 1 (Experimental): All participants
  Interventions: Other: Intervention 1: Electronic medical record (EMR)-based transitional care intervention

INTERVENTIONS:
Other: Intervention 1: Electronic medical record (EMR)-based transitional care intervention — Electronic delivery of enhanced discharge information to the ambulatory physician with plans for follow-up appointment, notice of any new medications, and recommendations for laboratory monitoring

SUMMARY:
The incidence of drug-induced injury is high in the ambulatory geriatric population, especially for elders with complex healthcare needs during high risk transitions to the ambulatory setting. In a previous study funded by the National Institute on Aging and the Agency for Healthcare Research and Quality [AHRQ] (AG 15979), the investigators determined that drug-related injuries occur at a rate of more than 50 per 1000-patient years in older adults in the ambulatory setting and that 28% are preventable. Independent risk factors for adverse drug events among older adults in the ambulatory setting included advanced age, multiple comorbid conditions, and the use of medications requiring close monitoring. In this project, Using HIT to Improve Transitions of Complex Elderly Patients from SNF to Home (1 R18 HS017817), the investigators are testing the use of an electronic medical record (EMR)-based transitional care intervention for complex elderly patients transitioning from subacute care in a skilled nursing facility (SNF) to the ambulatory setting. The growing trend for physicians and other healthcare providers to restrict their practices to single settings and not follow complex patients as they move between settings leaves older patients discharged from subacute care particularly vulnerable. This transition is uniquely challenging because of the complex healthcare needs of this population, who often require outpatient primary care physicians to coordinate with visiting nurses in order to manage complex medication regimens and fluctuating clinical status. To facilitate high-quality transitions from the subacute to the ambulatory setting and support interdisciplinary communication, the investigators will use the EMR to assure that physicians in the ambulatory setting receive key health information and alerts.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older,
* Member of the study site health plan,
* Received care from one of the study site's geriatricians during a SNF stay,
* Discharged from SNF to home.

Exclusion Criteria:

* Does not meet inclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 626 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of follow-up to an outpatient provider within 21 days of SNF discharge. | 1 year 3 months
Prevalence of appropriate monitoring for selected high risk medications at 30 days from the time of SNF discharge. | 1 year 3 months
Incidence of adverse drug events (ADEs) 45 days after discharge. | 1 year 3 months
Rate of SNF readmission and emergency department (ED) within 30 days of discharge. | 1 year 3 months

SECONDARY OUTCOMES:
Determine costs directly related to the development and installation of the HIT-based transitional care intervention | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Terry S Field, DSc, Principal Investigator — University of Massachusetts Medical School/Meyers Primary Care Institute
Locations (1):
- Fallon Clinic, Worcester, Massachusetts, United States